CLINICAL TRIAL: NCT01148758
Title: Open-label, Exploratory, Pharmacodynamic (PD) Dose-finding Study of Intravenous RO5323441 in Patients With Metastatic Treatment-refractory Colorectal and Ovarian Cancer
Brief Title: A Dose-finding Study of RO5323441 in Patients With Metastatic Treatment-Refractory Colorectal or Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP22909; 2009-016014-25
Record Dates: First submitted 2010-05-05; First posted 2010-06-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer, Ovarian Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms | interventions — TB-403

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5323441

INTERVENTIONS:
Drug: RO5323441 — cohorts receiving multiple doses iv

SUMMARY:
This exploratory, open label study will assess the the dose-effect relationship, efficacy and safety of RO5323441 in patients with metastatic treatment-refractory colorectal or ovarian cancer. Cohorts of patients will receive doses of intravenous RO5323441 in the range of 25mg to 3g every 1 or 2 weeks and will undergo serial dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) assessments. In the absence of disease progression and unacceptable toxicity, patients may continue to receive their maximum dose of RO5323441 for a core treatment phase of up to a total of 6 months. Treatment with RO5323441 can be extended at the investigator's discretion until disease progression or unacceptable toxicity occurs. Target sample size is <100.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=19 years of age
* metastatic or unresectable colorectal or ovarian cancer refractory to, or unsuitable for standard therapy
* presence of tumor lesions suitable for DCE-MRI evaluation
* WHO performance status 0-1
* adequate bone marrow, liver and renal function

Exclusion Criteria:

* patient unsuitable for MRI scanning (e.g. metal implants, pacemaker, claustrophobia, hypersensitivity to DCE-MRI contrast material)
* brain metastases
* clinically significant ascites
* active bleeding, bleeding diathesis, oral anti-vitamin K medication (other than low dose coumarin) or history of coagulation disorders
* radiation therapy within 3 weeks, or anti-neoplastic therapy <30 days prior to first dose of study drug
* chronic therapy with systemic steroids or another immunosuppressive agent <2 weeks prior to first dose of study drug
* treated with bevacizumab in last regimen of systemic therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
RO5323441 concentration - pharmacodynamic effect relationship using DCE-MRI | up to 19.5 months

SECONDARY OUTCOMES:
Feasibility of within-patient dose escalation | from baseline to Day 127 (+/-3)
Additional DCE-MRI effects (time-course of DCE-MRI effects, test-retest reproducibility) | up to 19.5 months
Candidate biomarkers associated with PD effect of RO5323441 | up to 19.5 months
Pharmacokinetics: maximum and trough concentrations of RO5323441 | up to 19.5 months
Safety and tolerability: Adverse events, vital signs, laboratory parameters | up to 19.5 months
Efficacy: ORR, duration of response, progression-free survival according to RECIST criteria, CTI/MRI assessments | up to 19.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Leuven, Belgium
- Barcelona, Barcelona, Spain
- Manchester, United Kingdom